CLINICAL TRIAL: NCT05837897
Title: A Phase 3, Multicenter, Randomized, Parallel-Group, Double-blind, Placebo-Controlled Induction Study Followed by an Open-label Extension Period to Evaluate the Efficacy and Safety of Intravenous Vedolizumab (300 mg) Infusion Treatment in Subjects in China With Moderately to Severely Active Crohn's Disease
Brief Title: A Study of Vedolizumab in Adult Participants With Moderate to Severe Crohn's Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vedolizumab-3040
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Crohn's Disease
Keywords: Drug therapy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Induction Period: Vedolizumab 300 mg (Experimental): Participants will receive vedolizumab 300 mg IV infusion on Days 1,15, and 43 (Weeks 0, 2, and 6) in the 14-week Induction Period.
  Interventions: Drug: Vedolizumab IV
- Induction Period: Placebo (Placebo Comparator): Participants will receive vedolizumab placebo-matching IV, infusion on Days 1,15, and 43 (Weeks 0, 2, and 6) in the 14-week Induction Period.
  Interventions: Drug: Placebo
- Open-label Extension (OLE) Period: Vedolizumab 300 mg (Experimental): All participants completing the Week 14 visit, irrespective of their response status, will continue in the OLE without unblinding of their baseline treatment group and will receive vedolizumab 300 mg, IV infusion, Q8W, on Days 99, 155, 211, 267, 323, and 379 (Weeks 14, 22, 30, 38, 46 and 54). Starting from Day 127 (Week 18) until the end of OLE Period up to approximately 58 weeks, participants who are nonresponders or who have disease worsening are eligible to receive 300 mg vedolizumab Q4W.
  Interventions: Drug: Vedolizumab IV

INTERVENTIONS:
Drug: Vedolizumab IV — Vedolizumab IV infusion
  Arms: Induction Period: Vedolizumab 300 mg; Open-label Extension (OLE) Period: Vedolizumab 300 mg
Drug: Placebo — Vedolizumab placebo-matching IV infusion
  Arms: Induction Period: Placebo

SUMMARY:
This is a study to evaluate vedolizumab for injection (300 mg) as a safe and active treatment for Crohn's Disease in adults in China. Participants will receive an injection of Vedolizumab 300 mg at scheduled weeks 0, 2, and 6, and starting at week 14, every 8 weeks over 58 weeks or starting at week 18, every 4 weeks over 54 weeks. There will be up to 20 study visits over 58 weeks to complete assessments.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. Vedolizumab will be administered as an intravenous (IV) infusion in Chinese participants. This study will investigate the efficacy and safety of vedolizumab IV in participants with moderately to severely active Crohn's Disease (CD).

The study will enroll approximately 408 patients. Participants will be randomized into 2:1 in the Induction Period to receive:

* Vedolizumab IV 300 mg
* Placebo

All participants completing the Week 14 visit, irrespective of their response status, will continue in the OLE without unblinding of their baseline treatment group and will receive 300 mg vedolizumab once every 8 weeks (Q8W) starting from Week 14. Starting at Week 18 and throughout the remainder of the OLE, participants who are nonresponders or who have disease worsening based on the assessment by visit every 4 weeks, are eligible to receive 300 mg vedolizumab once every 4 weeks (Q4W).

This multi-center trial will be conducted in China. The overall time participants will be in this study is approximately 58 weeks. Participants will make a final safety follow-up visit at 18 weeks after the last dose of study drug. Participants will also be followed-up for a long-term follow-up safety survey after completion of or early termination from study via telephone, 6 months after last dose of study drug.

ELIGIBILITY:
Inclusion criteria:

1. The participant has a diagnosis of CD established at least 3 months before screening by clinical and endoscopic evidence corroborated by a histopathology report. Cases of CD established at least 6 months before randomization for which a histopathology report is not available will be considered based on the weight of evidence supporting the diagnosis and excluding other potential diagnoses, and must be discussed with the sponsor on a case-by-case basis before randomization.
2. The participant has moderately to severely active CD as determined by a 2-component patient-reported outcome (PRO2) score of 14 to 34 points and a Simple Endoscopic Score for Crohn's Disease (SES-CD) score of ≥6 (or ≥4 in cases of isolated ileitis) on screening ileocolonoscopy.
3. The participant has CD involvement of the ileum and/or colon, at a minimum.
4. A participant with extensive colitis or pancolitis of >8 years duration or limited colitis of >12 years duration must have documented evidence that a surveillance colonoscopy was performed within 12 months before initial screening (may be performed during screening if not performed in previous 12 months).
5. A participant with a family history of colorectal cancer, personal history of increased colorectal cancer risk, age >50 years, or other known risk factor must be up-to-date on colorectal cancer surveillance (may be performed during screening).
6. The participant has demonstrated an inadequate response to, loss of response to, or intolerance of at least 1 of the following agents as defined below:

   * Corticosteroids.
   * Immunomodulators.
   * TNF-α antagonists.

Exclusion Criteria:

I. Gastrointestinal (GI) Exclusion Criteria:

1. The participant has evidence of abdominal abscess at the initial screening visit.
2. The participant has had extensive colonic resection, subtotal or total colectomy.
3. The participant has a history of >3 small bowel resections or diagnosis of short bowel syndrome.
4. The participant has received tube feeding, defined formula diets, or parenteral alimentation within 21 days before administration of the first dose of study drug.
5. The participant has had ileostomy, colostomy, known fixed symptomatic stenosis of the intestine, or evidence of fixed stenosis, or small bowel stenosis with prestenotic dilation.
6. Within 30 days before randomization, the participant has received any of the following for the treatment of underlying disease:

   * Nonbiologic therapies (eg, cyclosporine, thalidomide) other than those specifically listed in the Permitted Medications and Treatments section.
   * An approved or investigational nonbiologic therapy in an investigational protocol.
7. The participant has received traditional Chinese medication (TCMs) within 30 days before randomization.
8. The participant has had previous exposure to approved or investigational anti-integrins including, but not limited to natalizumab, efalizumab, etrolizumab, or abrilumab (AMG-181), or mucosal vascular addressin cell adhesion molecule 1 (MAdCAM-1) antagonists, or rituximab.
9. The participant has had previous exposure to vedolizumab.
10. The participant has used topical (rectal) treatment with 5-aminosalicylic acid (5-ASA), corticosteroid enemas/suppositories or traditional Chinese medications for CD treatment within 2 weeks of the administration of the first dose of study drug.
11. The participant requires currently or is anticipated to require surgical intervention for CD during the study.
12. The participant has a history or evidence of adenomatous colonic polyps that have not been removed.
13. The participant has a history or evidence of colonic mucosal dysplasia including low or high-grade dysplasia, as well as indeterminate for dysplasia.

    II. Infectious Disease Exclusion Criteria
14. The participant has evidence of active infection during the screening period.
15. The participant has evidence of treatment for Clostridioides difficile (C difficile) infection or other intestinal pathogen within, 28 days before first dose of study drug.
16. The participant has chronic hepatitis B virus (HBV) infection or chronic hepatitis C virus (HCV) infection.
17. The participant has active or latent tuberculosis (TB).
18. The participant has any identified congenital or acquired immunodeficiency (eg, common variable immunodeficiency, human immunodeficiency virus [HIV] infection, organ transplantation).
19. The participants has received any live vaccinations within 30 days before screening.
20. The participant has a clinically significant active infection (eg, pneumonia, pyelonephritis, or coronavirus disease 2019 [COVID-19]) within 30 days before screening or during screening, or has an ongoing chronic infection or any ongoing COVID-19-related symptom(s), if previously diagnosed as having COVID-19.

    III. General Exclusion Criteria
21. The participant has had any surgical procedure requiring general anesthesia within 30 days before enrollment or is planning to undergo major surgery during the study period.
22. The participant has any history of malignancy, except for the following: (a) adequately-treated nonmetastatic basal cell skin cancer; (b) squamous cell skin cancer that has been adequately treated and has not recurred for at least 1 year before randomization; and (c) history of cervical carcinoma in situ that has been adequately treated and has not recurred for at least 3 years before randomization. Participants with remote history of malignancy (eg, >10 years since completion of curative therapy without recurrence) will be considered based on the nature of the malignancy and the therapy received and must be discussed with the sponsor on a case-by-case basis before randomization.
23. The participant has a history of any major neurological disorders, including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2030-03-08 (Estimated); Study Completion 2031-05-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Clinical Response at Week 14 | Up to Week 14
  Clinical response is defined as ≥8 point decrease in 2-component patient-reported outcome (PRO2) score from baseline. The PRO2 is constituted by abdominal pain and number of liquid stools components of the Crohn's Disease Activity Index (CDAI). The PRO-2 score is the sum of the abdominal pain and stool frequency subscores of the CDAI score. The average daily number of liquid or very soft stools and abdominal pain score (with 0 indicating no pain and 3 indicating severe pain) are weighted according to the CDAI multiplication factors (2 for stool frequency and 5 for abdominal pain).

SECONDARY OUTCOMES:
Percentage of Participants Achieving Clinical Remission at Week 14 | Up to Week 14
  Clinical remission is defined as PRO2 score <8 from baseline. The PRO2 is comprised of the stool frequency and abdominal pain components of the CDAI. The PRO-2 score is the sum of the abdominal pain and stool frequency subscores of the CDAI score. The average daily number of liquid or very soft stools and abdominal pain score (with 0 indicating no pain and 3 indicating severe pain) are weighted according to the CDAI multiplication factors (2 for stool frequency and 5 for abdominal pain).
Percentage of Participants Achieving Endoscopic Response at Week 14 | Up to Week 14
  Endoscopic response is defined as Simple Endoscopic Score for Crohn's Disease (SES-CD) reduction by ≥50%. The SES-CD evaluates 4 endoscopic variables (ulcer size, percentage of the surface area that is ulcerated, percentage of the surface area affected, and presence and type of narrowings in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable is sum of values obtained for each segment. The SES-CD total is the sum of the 4 endoscopic variable scores from 0 to 60, where higher scores indicate more severe disease.
Percentage of Participants Achieving Both Clinical Response and Endoscopic Response at Week 14 | Up to Week 14
  Clinical response:≥8 point decrease in PRO2 score from baseline. Endoscopic response:SES-CD reduction by ≥50%.PRO2:number of liquid stools and abdominal pain components of the CDAI. PRO-2 score:sum of the abdominal pain and stool frequency subscores of the CDAI score.Average daily number of liquid or very soft stools and abdominal pain score (0=no pain and 3=severe pain) are weighted according to the CDAI multiplication factors (2= stool frequency;5= abdominal pain).Negative change indicates clinical response achieved.SES-CD evaluates 4 endoscopic variables (ulcer size, percentage of the surface area that is ulcerated, percentage of the surface area affected, and presence of narrowings) in 5 colonic segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum).Score for each endoscopic variable=sum of values obtained for each segment.SES-CD total=sum of the 4 endoscopic variable scores from 0 to 60, where higher scores=more severe disease.
Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs) and AEs Leading to Discontinuation | From first dose up to 18 weeks after the final dose of vedolizumab (Up to approximately 78 weeks)
  AE:any untoward medical occurrence in clinical investigation participants administered a drug;it does not necessarily have to have causal relationship with treatment.SAE:any untoward medical occurrence that:1)results in death,2)is life-threatening,3)requires inpatient hospitalization or prolongation of existing hospitalization,4)results in persistent or significant disability/incapacity,5)leads to a congenital anomaly/birth defect in offspring of participant or6)is medically important event that satisfies any of following:a)May require intervention to prevent items 1 through 5 above.b)May expose participant to danger,even though event is not immediately life threatening or fatal or does not result in hospitalization.AESI:serious infections,opportunistic infections such as progressive multifocal leukoencephalopathy(PML);liver injury;malignancies;infusion-related reactions,injection site reactions,systemic reactions,and hypersensitivity.
Percentage of Participants With Abnormal Change from Baseline in Vital Sign Values | From first dose up to 18 weeks after the final dose of vedolizumab (Up to approximately 78 weeks)
  Vital signs assessment will include body temperature, respiratory rate, blood pressure, and pulse (beats per minute). Abnormal values will be determined by the investigator.
Percentage of Participants With Abnormal Change from Baseline in Laboratory Values | From first dose up to 18 weeks after the final dose of vedolizumab (Up to approximately 78 weeks)
  Laboratory parameter assessment will include hematology, serum chemistry, and urinalysis. Abnormal values will be determined by the central lab.
Percentage of Participants With Abnormal Change from Baseline in Electrocardiogram (ECG) Values | From first dose up to 18 weeks after the final dose of vedolizumab (Up to approximately 78 weeks)
  The ECG results will be interpreted using 1 of the following categories: within normal limits, abnormal but not clinically significant, or abnormal and clinically significant. Abnormal values are determined by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (41):
- China (41):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Yijishan Hospital of Wannan Medical College, Wuhu, Anhui
  - Peking University First Hospital - Changqiao Campus, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University - Main, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - The University of Hong Kong - Shenzhen Hospital, Shenzhen, Guangdong
  - The Fifth Affiliated Hospital Sun Yat-Sen University, Zhuhai, Guangdong
  - The Second Hospital of Hebei Medical University - Main, Shijiazhuang, Hebei
  - The 2nd Affliated Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - Nanyang First People's Hospital, Nanyang, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University - Main Campus, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Changzhou No.2 People's Hospital - Yanling Campus, Changzhou, Jiangsu
  - Zhongda Hospital, Affiliated to Southeast University, Nanjing, Jiangsu
  - Changshu No.2 People's Hospital, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University - Donghu Campus, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University - Nanhu Campus, Shenyang, Liaoning
  - People's Hospital of Ningxia Hui Aotonomous Region, Yinchuan, Ningxia
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital - Main, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine - Qingchun Campus - PPDS, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Ningbo University - Fangqiao Campus, Ningbo, Zhejiang
  - People's Hospital of Quzhou, Quzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province - Main, Taizhou, Zhejiang
  - The First People's Hospital of Wenling, Taizhou, Zhejiang
  - The 1st Affiliated Hospital of Wenzhou Medical University - Nanbaixiang Campus, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/0b462a4eb07d47f4?idFilter=%5B%22Vedolizumab-3040%22%5D